CLINICAL TRIAL: NCT04620616
Title: A Randomized, Open-Label, Multi-Center, Cross-Over Study of Adult Electronic Nicotine Delivery Systems (ENDS) Consumers to Assess Nicotine Uptake, Measures of Abuse Liability, and Puffing Topography With RELX Infinity ENDS
Brief Title: Nicotine Uptake, Measures of Abuse Liability, and Puffing Topography With Use of RELX ENDS Products by ENDS Consumers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheerain HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RELX-002
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Electronic Cigarette Use
Keywords: Electronic Nicotine Delivery System; Nicotine; Pharmacokinetics; Abuse Liability; Topography; E-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product Use Sequence 1 (Experimental): Products use sequence:
  Period 1 - RELX ENDS tobacco flavor Period 2 - RELX ENDS menthol flavor Period 3 - Usual Brand ENDS
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS
- Product Use Sequence 2 (Experimental): Products use sequence:
  Period 1 - RELX ENDS menthol flavor Period 2 - Usual Brand ENDS Period 3 - RELX ENDS tobacco flavor
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS
- Product Use Sequence 3 (Experimental): Products use sequence:
  Period 1 - Usual Brand ENDS Period 2 - RELX ENDS tobacco flavor Period 3 - RELX ENDS menthol flavor
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS
- Product Use Sequence 4 (Experimental): Products use sequence:
  Period 1 - Usual Brand ENDS Period 2 - RELX ENDS menthol flavor Period 3 - RELX ENDS tobacco flavor
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS
- Product Use Sequence 5 (Experimental): Products use sequence:
  Period 1 - RELX ENDS tobacco flavor Period 2 - Usual Brand ENDS Period 3 - RELX ENDS menthol flavor
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS
- Product Use Sequence 6 (Experimental): Products use sequence:
  Period 1 - RELX ENDS menthol flavor Period 2 - RELX ENDS tobacco flavor Period 3 - Usual Brand ENDS
  Interventions: Other: RELX ENDS Tobacco Flavor; Other: RELX ENDS Menthol Flavor; Other: Subject Usual Brand ENDS

INTERVENTIONS:
Other: RELX ENDS Tobacco Flavor — Ad libitum use of the RELX ENDS tobacco flavor product during 8-hour and 5-minute use sessions
Other: RELX ENDS Menthol Flavor — Ad libitum use of the RELX ENDS tobacco flavor product during 8-hour and 5-minute use sessions
Other: Subject Usual Brand ENDS — Ad libitum use of the usual brand product during 8-hour and 5-minute use sessions

SUMMARY:
This study is being conducted to evaluate nicotine uptake, the potential abuse liability, and puffing topography associated with the use of an electronic nicotine delivery system (ENDS) with tobacco- and menthol-flavored e-liquids in current ENDS consumers.

ELIGIBILITY:
Inclusion Criteria:

1. Provides voluntary consent to participate in the study as documented on the signed informed consent form (ICF).
2. Is 22 to 59 years of age, inclusive, at the time of consent.
3. Has been a daily ENDS consumer for at least 3 months prior to Screening and through Check-in. Brief periods of abstinence (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where vaping was prohibited) ≥ 30 days prior to Screening will be permitted at the discretion of an Investigator.
4. Reports weekly use of at least 3 mL of e-liquid from an ENDS product at Screening.
5. Has a urine cotinine concentration ≥ of 200 ng/mL at Screening and Check-in.
6. Has an exhaled carbon monoxide (ECO) concentration < 10 ppm at Check-in.
7. If female, must meet one of the following criteria:

   If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first product use, during the study, and for at least 30 days after the last product use. An acceptable method of contraception includes one of the following: abstinence from heterosexual intercourse, hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch), intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g. condom and spermicide) during the study and for at least 30 days after the last product use.

   If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels (≥ 40 mIU/mL).
8. Is willing to comply with the requirements of the study.

Exclusion Criteria:

1. Has a history or presence of clinically significant uncontrolled gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that would jeopardize the safety of the subject or impact the validity of the study results.
2. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results.
3. Has a positive test for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen, or Hepatitis C Antibody.
4. Has had an acute illness (e.g., upper respiratory infection, viral infection) within 14 days prior to Check-in.
5. Has a fever (> 100.5°F) at Screening or Check-in.
6. Has a positive COVID-19 test during the screening period, prior to Check-in.
7. Has a body mass index greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening.
8. Has a history of drug or alcohol abuse within 12 months of Screening.
9. Has a systolic BP < 90 mmHg or > 150 mmHg, diastolic BP < 40 mmHg or > 95 mmHg, or HR < 40 bpm or > 99 bpm at Screening.
10. Is allergic to or intolerant of components of the product e-liquid, including but not limited to, menthol, propylene glycol or glycerin.
11. Is unable to use the CReSS topography device with the vaping device during the training session on Day -1.
12. Has an estimated creatinine clearance < 70 mL/minute (using the Cockcroft Gault equation) at Screening.
13. Has a positive urine drug or alcohol test at Screening or Check-in. A positive test result for cannabinoids may be permitted if the result to the cannabis intoxication evaluation is negative at Check-in.
14. If female, has a positive pregnancy test, is breastfeeding or lactating, or intends to become pregnant from Screening through Day 5.
15. Has been treated for depression, diabetes, asthma, emphysema, or chronic obstructive pulmonary disease within 12 months of Check-in.
16. Has previously been diagnosed with any form of cancer, except for basal cell or squamous epithelial carcinomas of the skin that have been resected.
17. Has used medications known to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, desipramine, isoniazid, ketoconazole, miconazole, phenobarbital, rifampin, tranylcypromine, methoxsalen) within 6 weeks prior to Check-in.
18. Has used a product containing pseudoephedrine within 48 hours prior to Check-in.
19. Has used any other tobacco- or nicotine-containing products other than closed-system ENDS products (e.g., open-system ENDS, cigarettes, cigars, pipes, snuff, pouches, chewing tobacco, nicotine inhalers, nicotine patches, nicotine sprays, nicotine lozenges, or nicotine gum) within 7 days of Check-in.
20. Has used any products for the purpose of smoking/vaping cessation, including, but not limited to, nicotine replacement therapies, varenicline (Chantix), or bupropion (Zyban) from 30 days prior to Screening through Check-in.
21. Is a self-reported puffer (i.e., draws aerosol from the ENDS into the mouth and throat but does not inhale).
22. Is postponing a planned vaping quit attempt in order to participate in the study.
23. Has donated plasma within 7 days prior to Check-in.
24. Has provided a whole blood donation, had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Check-in.
25. Has participated in a previous clinical study for a tobacco product or an investigational drug, device, or biologic, within 30 days or 5 times the half-life of the product (whichever is longer) prior to Check-in.
26. Is or has a first-degree relative (e.g., spouse, parent, sibling, child) who is a current or former employee of a tobacco or ENDS manufacturer or is a named party or class representative in litigation with the tobacco or ENDS industry.
27. Is or has a first-degree relative (e.g., spouse, parent, sibling, child) who is a current employee of the clinic site(s).
28. Is or has a first-degree relative (e.g., spouse, parent, sibling, child) who is a current employee of the Sponsor.
29. Has previously been withdrawn from or has completed this study.
30. In the opinion of an Investigator, the subject should not participate in this study.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Nicotine uptake | 120 minutes
  PK Session baseline-adjusted maximum plasma nicotine concentration [Cmax]
Nicotine uptake | 120 minutes
  PK Session baseline-adjusted area under the nicotine concentration-time curve [AUC(0-120)]

SECONDARY OUTCOMES:
Nicotine uptake - PK Session | 15 minutes
  PK Session baseline-adjusted area under the nicotine concentration-time curve [AUC(0-15)]
Nicotine uptake - PK Session | 120 minutes
  PK Session time of the maximum post-baseline nicotine concentration [Tmax]
Nicotine uptake - Ad Libitum Session | 480 minutes
  Ad Libitum Session baseline-adjusted area under the nicotine concentration-time curve [AUC(0-480)]
Subject effects as measured by the Modified Product Evaluation Scale | 480 minutes
  Subjective product assessments during the Ad Libitum Session as measured by responses to the Modified Product Evaluation Scale (scale range of 1 [not at all] to 7 [extremely])
Subject effects as measured by the Future Intent to Use questionnaire | 480 minutes
  Subjective product assessments during the Ad Libitum Session as measured by responses to the Future Intent to Use questionnaire (visual analog scale range of "Definitely Would Not" to "Definitely Would")
Subject effects as measured by the Urge to Vape questionnaire | 120 minutes
  Subjective product assessments during the PK Session as measured by responses to the Urge to Vape questionnaire (visual analog scale range of "Not at All" to "Extreme")
Subject effects as measured by the Product Liking questionnaire | 120 minutes
  Subjective product assessments during the PK Session as measured by responses to the Product Liking questionnaire (visual analog scale range of "Not at All" to "Extremely")
Physiologic effects as measured by heart rate | 480 minutes
  Heart rate measurements during the Ad Libitum Session
Physiologic effects as measured by heart rate | 120 minutes
  Heart rate measurements during the PK Session
Physiologic effects as measured by blood pressure | 480 minutes
  Blood pressure measurements during the Ad Libitum Session
Physiologic effects as measured by blood pressure | 120 minutes
  Blood pressure measurements during the PK Session
Study product use | 480 minutes
  Change in weight of study products during the Ad Libitum Session
Study product use | 480 minutes
  Number of requests to use the study products during the Ad Libitum Session
Study product use | 60 minutes
  Number of puffs taken from the study products during the Ad Libitum Session topography assessment
Study product use | 60 minutes
  Duration of puffs taken from the study products during the Ad Libitum Session topography assessment
Study product use | 60 minutes
  Volume of puffs taken from the study products during the Ad Libitum Session topography assessment
Study product use | 60 minutes
  Flow rate of puffs taken from the study products during the Ad Libitum Session topography assessment
Study product use | 60 minutes
  Inter-puff interval of puffs taken from the study products during the Ad Libitum Session topography assessment
Study product use | 5 minutes
  Change in weight of study products during the PK Session
Study product use | 5 minutes
  Number of puffs taken from the study products during the PK Session
Safety and tolerability | 24 hours
  Incidence of product-use emergent adverse events
Safety and tolerability | 24 hours
  Incidence of product malfunction or misuse

CONTACTS AND LOCATIONS:
Overall Officials: Donald Graff, PharmD, Study Director — Sponsor Representative
Locations (2):
- United States (2):
  - WCCT Global, Inc, Cypress, California
  - Altasciences Clinical Kansas, Inc, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No